CLINICAL TRIAL: NCT00205283
Title: Nelfinavir and M8 Drug-level Monitoring in HIV-1 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Agouron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2002-212
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — Nelfinavir

INTERVENTIONS:
Drug: Nelfinavir

SUMMARY:
The purpose of this study is to assess the impact of prospective drug level monitoring and dose-adjustment of nelfinavir (NFV) on the clinical and virologic outcomes in a group of HIV-infected patients who have achieved virologic success while receiving a nelfinavir containing highly active antiretroviral therapy (HAART) regimen.

ELIGIBILITY:
Inclusion Criteria:

* Antiretroviral naive or currently taking a nelfinavir containing HAART regimen where nelfinavir is the first protease inhibitor
* Patients willing to comply with the protocol
* Age greater than or equal to 18 years
* Virologically successful if already on an established regimen

Exclusion Criteria:

* Prior use of a protease inhibitor exclusive of nelfinavir
* Required use or concomitant use of drugs that may interact with or are contraindicated with nelfinavir
* Use of immunomodulators or vaccines for HIV disease
* Intercurrent illness at the time of enrollment that, in the clinician's judgement, could influence the HIV RNA concentration
* Baseline ALT levels greater than five times the upper limit of normal

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-08; Primary Completion 2005-08-01 (Actual); Study Completion 2005-08-01 (Actual)

PRIMARY OUTCOMES:
Virologic response
Nelfinavir pharmacokinetics

SECONDARY OUTCOMES:
Impact of nelfinavir and M8 pharmacokinetics on virologic response

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Urban, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States